CLINICAL TRIAL: NCT05633238
Title: SSVEP and Distractor Processing During Visual Search in Healthy Adults
Brief Title: SSVEP and Distractor Processing During Visual Search
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lehigh University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 3R15EY030247-01A1 (NIH)
Record Dates: First submitted 2022-11-07; First posted 2022-12-01 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2023-10

CONDITIONS: Healthy
Keywords: attention; visual search

STUDY DESIGN:
Intervention Model Description: All participants receive each level of visual information (target or distractor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Within-Subjects Attentional Information (Experimental): Within-Subjects, all participants receive all interventions
  Interventions: Behavioral: Visual Search Information Type (target or distractor information)

INTERVENTIONS:
Behavioral: Visual Search Information Type (target or distractor information) — Participants will have information about targets, distractors, or neither in different blocks of the intervention.

SUMMARY:
In this line of research, the researchers are utilizing an EEG measure of repeated visual stimulation, the Steady-State Visually Evoked Potential (SSVEP) to examine processing of target and distractor information during visual search. This is a basic science study.

DETAILED DESCRIPTION:
The researchers are interested in how the brain responds to target and distractor information during visual search. The researchers will manipulate the information available to the research participants, and measure research participants brain responses to information matching target or distractor features utilizing an EEG measure of repeated visual stimulation, the Steady-State Visually Evoked Potential (SSVEP).

ELIGIBILITY:
Inclusion Criteria:

* normal or corrected to normal visual acuity, normal color vision

Exclusion Criteria:

* history of neurological disorders

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Steady-State Visually Evoked Response (SSVEP) | One day (during testing)
  Brain response to visual stimuli flashing at a pre-defined frequency
Button Press Reaction Time | One day (during testing)
  Speed to respond correctly to the target- after participant finds the target shape on a computer screen, they press a button to indicate what shape they see
Button Press Accuracy | One day (during testing)
  Accuracy of responses to target item (% correct)- the researchers will measure whether the participants presses the correct button which corresponds to the target shape presented on the computer screen or the incorrect button

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Carlisle, PhD, Principal Investigator — Lehigh University
Locations (1):
- Lehigh University, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers plan to share anonymized subject data on Open Science Framework.
Supporting Information: Study Protocol, SAP
Time Frame: Upon publication.
Access Criteria: Open Science Framework internet access.